CLINICAL TRIAL: NCT01749267
Title: Clinical and Digital Subtraction Radiography Evaluation of Partial Caries Removal in Primary Teeth
Brief Title: Digital Subtraction Radiography Evaluation of SMART Restoration With Partial Caries Removal in Primary Teeth
Acronym: DSR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Faculty of Dentistry
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2010-09

CONDITIONS: Dental Caries Extending Into Dentine
Keywords: dentin remineralization; caries regression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- partial caries removal (Experimental): partial caries removal only at enamel dentin junction (EDJ) without carious tissue removal at the pulpal site
  Interventions: Procedure: partial caries removal only at enamel dentin junction.

INTERVENTIONS:
Procedure: partial caries removal only at enamel dentin junction. — Partial caries removal only at enamel dentin junction (EDJ) without carious dentin removal at the pulpal site and restoration with glass ionomer cement(SMART restoration)

SUMMARY:
The objective of this study was to analyze the radiographic density of digital subtraction radiographs after SMART restoration with partial caries removal in primary molars at 6 and 12 months.

DETAILED DESCRIPTION:
In management of deep caries in primary teeth, the partial caries removal approach favored the arrest of dentin carious lesions, reduced cariogenic micro-organisms and the risk of pulp exposure. The carious tissue at the lateral walls of the cavity at the enamel dentin junction (EDJ) was removed by a spoon excavator without carious tissue removal at the pulpal site. After caries removal, restoration using glass ionomer cement (GIC)(GC Fuji IX™GP extra) was completed. Such an approach is called SMART restoration. The serial radiographs of each restoration consisted of three radiographs; immediately after restoration, at the 6-month follow-up and at the 12-month follow-ups. Digital subtraction radiography(DSR) was used to evaluate dentin remineralization following partial caries removal. Image-Pro Plus software was used to evaluate DSR. For evaluating the changes in DSR, areas with increase density show higher radiopacity, whereas areas with decreased density show higher radiolucency. The 6-month and 12-month follow-up radiographs were subtracted from the baseline radiograph.

ELIGIBILITY:
Inclusion Criteria:

* Presence of teeth with dentinal caries limited to the occlusal and proximal surfaces without clinical signs and symptoms of irreversible pulpitis (spontaneous pain, sinus opening, or abnormal tooth mobility
* The radiographic examination showing dental caries involving not less than half of the dentin without any pathologic findings (external root resorption, internal root resorption, abnormality of root resorption, or radiolucency area at furcation /periapical regions).

Exclusion Criteria:

* Teeth with caries exposure to pulp

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2010-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
dentin remineralization | 12 months
  Dentin remineralization was evaluated using Digital subtraction radiography (DSR).

CONTACTS AND LOCATIONS:
Overall Officials: Araya Phonghanyudh, PhD, Study Director
Locations (1):
- Mahidol University, Bangkok, Bangkok, Thailand

REFERENCES:
- [Background] Phonghanyudh A, Phantumvanit P, Songpaisan Y, Petersen PE. Clinical evaluation of three caries removal approaches in primary teeth: a randomised controlled trial. Community Dent Health. 2012 Jun;29(2):173-8. PMID 22779380
- See also: Clink here for more information about this study:http://www.ncbi.nlm.nih.gov/pubmed?term=clinical evaluation of three caries removal approaches in primary teeth — http://www.ncbi.nlm.nih.gov/pubmed/22779380